CLINICAL TRIAL: NCT02792465
Title: An Open Label, Dose Escalation, Safety, and Pharmacokinetic Study of CFI-402257 Administered Orally to Patients With Advanced Solid Tumors
Brief Title: A Study of Investigational Drug CFI-402257 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFI-402257-CL-001
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Cancers; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CFI-402257; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Cohort A: Patients with advanced cancer. Treatment: Daily dose of 168 mg of CFI 402257.
  Cohort B: Patients with advanced breast cancer Treatment: Daily dose of 168 mg of CFI 402257.
  Cohort C: Patients with breast cancer tested positive for ER and/or PR, and HER2-negative. Treatment: Daily dose of 168 mg of CFI 402257 + Fulvestrant (standard hormonal treatment) on Day 1 and 15 of each 28 day cycle
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental): CFI-402257 capsules will be taken orally, once a day, every day.
  Interventions: Drug: CFI-402257
- Cohort B (Experimental): CFI-402257 capsules will be taken orally, once a day, every day.
  Interventions: Drug: CFI-402257
- Cohort C (Experimental): CFI-402257 capsules will be taken orally, once a day, every day + Fulvestrant injection on day 1 and day 15 of every 28 day cycle
  Interventions: Drug: CFI-402257; Drug: Fulvestrant

INTERVENTIONS:
Drug: CFI-402257
Drug: Fulvestrant
  Arms: Cohort C

SUMMARY:
This is a phase 1 study of investigational agent CFI-402257 in patients with advanced cancer. The purpose of this study is to see how safe and tolerable CFI-402257 is in cancer patients as well as the pharmacokinetics (PK). This study is the first time that CFI-402257 is given to humans.

DETAILED DESCRIPTION:
CFI-402257 is an oral drug that blocks TTK protein kinase (also known as Monopolar spindle 1 [Mps1]) activity. TTK is a protein that is important in regulating cell growth, and cell death, and ensuring proper division. Many tumors are shown to make too much TTK. When there is too much TTK produced, it is believed to contribute to uncontrolled cancer cell growth and division leading to additional mutations in cancer cells. Therefore, it is believed that blocking this protein from working will lead to cancer cell death, stopping tumors from growing or shrinking them.

This study has two parts: dose escalation and dose expansion.

The dose escalation part tested different dose levels of study drug in groups of patients to find the highest dose of study drug that can be given safely to patients (called maximum tolerated dose or MTD). This part of the study is now complete.

The expansion part will further assess the safety, tolerability, and PK of the MTD found in the escalation part of the study in additional group of patients.

ELIGIBILITY:
Inclusion Criteria - Cohort A:

* Have histological or cytological proof of advanced cancer that has progressed and for which there is no further standard anticancer therapy available in the opinion of the Investigator.
* Patients must have measurable disease as per RECIST v 1.1 guidelines.
* Patients must be ≥18 years of age.
* Have clinically acceptable laboratory screening results (i.e., clinical chemistry, hematology, and urinalysis) within certain limits.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Be able to swallow oral medications.
* Have a life expectancy of greater than 3 months.
* Women and men of child-producing potential must agree to use highly effective means of contraception for a specified period.
* A negative serum pregnancy test for women of childbearing potential.
* Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, provide archived tissue if available for biomarker studies, provide a blood sample for genetic testing and agree to return for the required assessments.

Inclusion Criteria - Cohort B:

* Have histologically and/or cytologically confirmed diagnosis of breast cancer that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists.
* Patients must have had at least 1 but not more than 4 prior lines of cytotoxic chemotherapy for breast cancer in the advanced/metastatic setting, and must have had prior treatment with an anthracycline and a taxane (unless contraindicated) in either the neo/adjuvant or metastatic setting.
* Patients must have measurable disease as per RECIST v 1.1 guidelines.
* Patients must be female.
* Patients must be ≥18 years of age.
* Have clinically acceptable laboratory screening results (i.e., clinical chemistry, hematology, and urinalysis) within certain limits.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Be able to swallow oral medications.
* Have a life expectancy of greater than 3 months.
* Women of child-producing potential must agree to use highly effective means of contraception for a specified period.
* A negative serum pregnancy test for women of childbearing potential.
* Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, provide archived tissue if available for biomarker studies, provide a blood sample for genetic testing and agree to return for the required assessments.

Inclusion criteria - Cohort C:

* Have histological or cytological confirmed diagnosis of breast cancer positive for ER and/or PR and negative for HER2 by ASCO/CAP criteria, that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists.
* Patients must have had prior treatment with an aromatase inhibitor in combination with CDK4/6 inhibitor, for a duration of not less than 12 months prior to disease progression. Up to 1 line of cytotoxine chemotherapy in the metastatic setting is allowed.
* Patients must have measurable disease as per RECIST v 1.1 guidelines.
* Patients must be female.
* Patients must be ≥18 years of age.
* Patients are post-menopausal (including use of ovarian function suppression with LHRH agonist)
* Have clinically acceptable laboratory screening results (i.e., clinical chemistry, hematology, and urinalysis) within certain limits.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Be able to swallow oral medications.
* Have a life expectancy of greater than 3 months.
* Women of child-producing potential must agree to use highly effective means of contraception for a specified period.
* A negative serum pregnancy test for women of childbearing potential.
* Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, provide archived tissue if available for biomarker studies, provide a blood sample for genetic testing and agree to return for the required assessments.

Exclusion Criteria (all cohorts):

* Women who are pregnant or nursing.
* Have received radiotherapy (patients having limited field palliative radiotherapy less than 2 weeks), chemotherapy, biological therapy, or investigational treatment less than four weeks (six weeks for nitrosoureas or mitomycin C) prior to first dose of study drug or have not recovered from all acute toxicities from prior treatments and those deemed by the Investigator not to affect safety assessment.
* Patients who have received growth factors within 14 days prior to initiation of dosing of CFI-402257 or who will require ongoing treatment with growth factors throughout the duration of the trial.
* Have active, acute, or clinically significant chronic infections.
* Have uncontrolled severe hypertension.
* Have symptomatic congestive heart failure.
* Have active angina pectoris or recent myocardial infarction (within 6 months).
* Have chronic atrial fibrillation or QTc of greater than 470 msec.
* Have had major surgery within 21 days of starting therapy.
* Have additional uncontrolled serious medical or psychiatric illness.
* Have any medical condition that would impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled nausea or vomiting.
* Known central nervous system metastasis.
* Patients being treated with full dose warfarin are excluded.
* Patients being treated with the following drugs are excluded: Alfentanil, Pimozide, Cyclosporine, Quinidine, Digoxin, Sirolimus, Dihydroergotamine, Tacrolimus, Ergotamine, Warfarin, Fentanyl.
* Patient who have had prior treatment with a TTK/MPS1 inhibitor
* For Expanded Cohort C - have previously been treated with, or have a contraindication to treatment with fulvestrant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2016-11-11 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Highest dose level that does not lead to unacceptable toxicity in two or more patients in a dosing cohort | 2 years

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) graded according to NCI CTCAE v4.03 | 2 years
Treatment-emergent changes in vital signs | 2 years
Treatment-emergent changes in clinical laboratory tests from baseline values obtained prior to treatment | 2 years
Treatment-emergent changes in physical examinations, ECOG performance status, electrocardiograms (ECGs), at periodic intervals during the study and at End of Treatment | 2 years
Area under the plasma concentration-time curve (AUC) | 2 years
Elimination half-life (T½) | 2 years
Maximum plasma concentration (Cmax) | 2 years
Minimum plasma concentration (Cmin) | 2 years
Time when Cmax occurs (Tmax) | 2 years
Average plasma concentration at steady state (Cavg) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (3):
- Canada (3):
  - BC Cancer Agency, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No